CLINICAL TRIAL: NCT03580265
Title: Efficacy of Laser Acupuncture for Carpal Tunnel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Chuan-Chih Chen, Attending Physician of Department of Chinese Medicine, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TSGHIRB: 1-107-05-062
Record Dates: First submitted 2018-06-25; First posted 2018-07-09 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Six-sessions of laser acupuncture (Experimental): Laser acupuncture was given three times a week for 2 weeks.
  Interventions: Device: laser phototherapy device with low level laser
- Six-sessions of sham laser acupuncture (Sham Comparator): Sham laser acupuncture was given three times a week for 2 weeks.
  Interventions: Device: laser phototherapy device with low level laser

INTERVENTIONS:
Device: laser phototherapy device with low level laser — The wavelength of low level laser is 808nm and the power output of low level laser is 300mW.

SUMMARY:
The laser acupuncture is a new and potential intervention for the disease of peripheral nerve. The purpose of this study was to assess the effect of laser acupucnture therapy on carpal tunnel syndrome.

DETAILED DESCRIPTION:
Laser acupuncture is combined low level laser with acupuncture points. Investigators perform a prospective randomized, single-blinded study to investigate the efficacy of laser acupuncture in patients with carpal tunnel syndrome. Patients were randomized into intervention and control group. Participants in intervention group received six-sessions of laser acupuncture and six-sessions of sham laser acupuncture was given in control group. All participants used wrist splint at night. The evaluation was performed pretreatment as well as on the 2th, 4th, 8th and 12th week after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-80 year-old.
* Typical symptoms and signs of mild to moderate carpal tunnel syndrome, such as positive Tinel's sign numbness/tingling in at least 5th digits, and in whom the diagnosis was confirmed using an electrophysiological study.

Exclusion Criteria:

* Cancer
* Coagulopathy
* Pregnancy
* Inflammation status
* Patients who had conditions mimicking carpal tunnel syndrome, such as cervical radiculopathy, polyneuropathy, brachial plexopathy, thoracic outlet syndrome or who had previously undergone wrist surgery or steroid injection for carpal tunnel syndrome.
* There are tattoos, birthmarks and skin disorders over acupuncture points.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of severity of symptoms and functional status on 2th, 4th, 8th and 12th weeks after treatment by using Boston Carpal Tunnel Questionnaire (BCTQ). | baseline, 2th, 4th, 8th and 12th weeks after treatment
  The Boston Carpal Tunnel Questionnaire (BCTQ) is a disease-specific measure of self-reported symptom severity and functional status. One is the minimum score and five is the maximum score in each symptom severity scale (11 items). The total score range of symptom severity scale is 11 to 55. One is the minimum score and five is the maximum score in each functional status scale (8 items). The total score range of functional status scale is 8 to 40.
  Using the Boston Carpal Tunnel Questionnaire to measure the symptoms and functional status of carpal tunnel syndrome before treatment and multiple time frame after treatment.

SECONDARY OUTCOMES:
Change from baseline of pain on 2th, 4th, 8th and 12th weeks after treatment by using Visual analog scale (VAS). | baseline, 2th, 4th, 8th and 12th weeks after treatment
  The visual analog scale (VAS) is a measurement instrument that tries to measure the amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain. Zero is the minimum score of pain and ten is the maximum score of pain.
  Using Visual analog scale (VAS) to measure the pain induced by carpal tunnel syndrome before treatment and multiple time frame after treatment.
Change from baseline of electrophysiological study and sonography on 2th, 4th, 8th and 12th weeks by using electrophysiological and sonographical machine measurement. | baseline, 2th, 4th, 8th and 12th weeks after treatment
  Electrophysiological study and sonography according to the protocol reported by the American Academy of Neurology with SierraWave, Cadwell (USA).

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital National Defense Medical Center, Taipei, Neihu Dist., Taiwan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Naeser MA, Hahn KA, Lieberman BE, Branco KF. Carpal tunnel syndrome pain treated with low-level laser and microamperes transcutaneous electric nerve stimulation: A controlled study. Arch Phys Med Rehabil. 2002 Jul;83(7):978-88. doi: 10.1053/apmr.2002.33096. PMID 12098159
- [Background] Baxter GD, Bleakley C, McDonough S. Clinical effectiveness of laser acupuncture: a systematic review. J Acupunct Meridian Stud. 2008 Dec;1(2):65-82. doi: 10.1016/S2005-2901(09)60026-1. PMID 20633458
- [Background] Fusakul Y, Aranyavalai T, Saensri P, Thiengwittayaporn S. Low-level laser therapy with a wrist splint to treat carpal tunnel syndrome: a double-blinded randomized controlled trial. Lasers Med Sci. 2014 May;29(3):1279-87. doi: 10.1007/s10103-014-1527-2. Epub 2014 Jan 30. PMID 24477392
- [Background] Wu YT, Ho TY, Chou YC, Ke MJ, Li TY, Huang GS, Chen LC. Six-month efficacy of platelet-rich plasma for carpal tunnel syndrome: A prospective randomized, single-blind controlled trial. Sci Rep. 2017 Dec;7(1):94. doi: 10.1038/s41598-017-00224-6. Epub 2017 Mar 7. PMID 28273894
- [Derived] Chen CC, Wu YT, Su YC, Shen YP, Chen FP. Efficacy of laser acupuncture for carpal tunnel syndrome: A study protocol for a prospective double-blind randomized controlled trial. Medicine (Baltimore). 2019 Jul;98(30):e16516. doi: 10.1097/MD.0000000000016516. PMID 31348263